CLINICAL TRIAL: NCT04324047
Title: Cohort Multiple Randomized Controlled Trials Open-label of Immune Modulatory Drugs and Other Treatments in COVID-19 Patients
Acronym: CORIMUNO-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200375; 2020-001246-18 (EudraCT Number)
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective of the study is to determine which treatments (e.g. immune modulator drugs) have the most favorable benefit-risk in adult patients hospitalized with COVID-19 either diagnosed with moderate or severe pneumonia requiring no mechanical ventilation or critical pneumonia requiring mechanical ventilation.

The specific aims of this Covid19 cohort are to collect observational data at regular intervals on an ongoing basis in order to embed a series of randomized controlled trials evaluating a various set of interventions for patients with COVID-19 pneumonia. The study has a cohort multiple Randomized Controlled Trials (cmRCT) design.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen < 72 hours and/or CT Scan prior to randomization (Following typical radiological findings (ground glass abnormalities, and absence of lymphadenopathy, pleural effusion, pulmonary nodules, lung cavitation)
* Hospitalized patients
* Illness of any duration and severity (mild, moderate, severe, critical, see annexe 1), with symptoms (fever, cough, respiratory difficulties, shortness of breath), and at least one of the following:
* Radiographic infiltrates by imaging (CT scan)
* Clinical assessment (evidence of rales/crackles on exam or respiratory rate >25/min) AND SpO2≤94% on room air
* SpO2≤97 % with O2 > 5L/min or Respiratory rate>=30/min
* Requiring mechanical ventilation
* With any comorbidities (TBD such as acute kidney injury, cardiovascular condition, pulmonary disease, obesity, high blood pressure, diabetes, chronic kidney diseases, haematological diseases, sickle cell diseases, autoimmune and auto-inflammatory, pregnant women, HIV infected, etc)
* Male or female adult ≥ 18 years of age at time of enrolment
* Patients must be able and willing to comply with study visits and procedures.
* Patient agrees to the collection of oropharyngeal and nasal swabs and venous blood per protocol Written informed consent provided by the patient or alternatively by next-of-kin prior to any protocol-specific procedures.

Exclusion Criteria:

* Patients with any condition that the physician judges could be detrimental to the patient participating in this study; including any clinically important deviations from normal clinical laboratory values or concurrent medical conditions (active infection diseases such as severe bacterial infections, aspergillosis, tuberculosis, depending on the tested medication).
* Absence of Health Insurance
* Subject protected by law under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients with laboratory-confirmed SARS-CoV-2 infection
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2021-03-27 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 14 days
  Overall Survival
WHO progression scale COVID 19 | 14 days
  Uninfected; non viral RNA detected: 0 Asymptomatic; viral RNA detected: 1 Symptomatic; Independent: 2 Symptomatic; Assistance needed: 3 Hospitalized; No oxygen therapy: 4 Hospitalized; oxygen by mask or nasal prongs: 5 Hospitalized; oxygen by NIV or High flow: 6 Intubation and Mechanical ventilation, pO2/FIO2>=150 OR SpO2/FIO2>=200: 7 Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min): 8 Mechanical ventilation, pO2/FIO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR ECMO: 9 Dead: 10

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Kremlin Bictre APHP, Le Kremlin-Bicêtre, Île-de-France Region
  - Cochin Aphp, Paris, Île-de-France Region
  - Hegp Aphp, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lenoir O, Morin F, Walter-Petrich A, Resmini L, Zaidan M, Mahtal N, Ferlicot S, Puelles VG, Wanner N, Dang J, d'Izarny-Gargas T, Biermann J, Izar B, Baron S, Terrier B, Massy ZA, Essig M, Couturier A, May O, Belenfant X, Buob D, Brocheriou I, Izzedine H, Lombardi Y, Francois H, Moktefi A, Audard V, Sannier A, Daugas E, Jamme M, Henry G, Le Monnier de Gouville I, Marie C, Homyrda L, Verstuyft C, Tubiana S, Kafif O, Piquard V, Dougados M, Huber TB, Livrozet M, Hulot JS, Laouenan C, Ghosn J, Mentre F, Karras A, Yazdanpanah Y, Porcher R, Ravaud P, Caillat-Zucman S, Mariette X, Hermine O, Resche-Rigon M, Tharaux PL; CORIMUNO-19 collaborative group. Levels of circulating kidney injury markers and IL-10 identify non-critically ill patients with COVID-19 at risk of death. JCI Insight. 2026 Jan 23;11(2):e198244. doi: 10.1172/jci.insight.198244. eCollection 2026 Jan 23. PMID 41574613
- [Derived] Dal-Re R. COVID-19 drug research and the cohort multiple randomised controlled trial design. Eur Respir J. 2022 Sep 15;60(3):2200746. doi: 10.1183/13993003.00746-2022. Print 2022 Sep. PMID 35896204
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343